CLINICAL TRIAL: NCT04883411
Title: First-in-human Prospective Study to Assess the Safety and Efficacy of the CEM-Cage and CEM-Plate
Brief Title: CEM-Plate and CEM-Cage First-In-Human Use Efficacy Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ReVivo Medical, Corp. (Industry)
Collaborators: Albany Medical College (Other); The Cleveland Clinic (Other); IGEA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RM-21-001
Record Dates: First submitted 2021-05-05; First posted 2021-05-12 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain; Spondylosis; Spondylosis With Myelopathy; Spondylosis With Radiculopathy; Spondylosis With Radiculopathy Cervical Region; Intervertebral Disc Disorder Cervical
Keywords: Cervical Spondylosis; Cervical Myelopathy; Cervical Radiculopathy; Neck Pain
MeSH Terms: conditions — Neck Pain; Spondylosis; Radiculopathy

STUDY DESIGN:
Intervention Model Description: Prospective, first-in-human, multi-center, non-randomized, single arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment (Experimental): Two-Level ACDF with CEM-Plate Anterior Cervical Plating System and CEM-Cage Cervical Interbody System.
  Interventions: Device: CEM-Plate Anterior Cervical Plating System and CEM-Cage Cervical Interbody System

INTERVENTIONS:
Device: CEM-Plate Anterior Cervical Plating System and CEM-Cage Cervical Interbody System — Two-Level ACDF with CEM-Plate Anterior Cervical Plating System and CEM-Cage Cervical Interbody System

SUMMARY:
The study is a prospective, first-in-human, multi-center, non-randomized, single-arm study to assess the safety and efficacy of the CEM-Cage used with the CEM-Plate in patients who are appropriate candidates for a 2-level anterior cervical discectomy and fusion (ACDF). Fifty patients will be enrolled in the study and, after undergoing a 2-level ACDF, will be evaluated at 4 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months.

DETAILED DESCRIPTION:
The study is a prospective, first-in-human, multi-center, non-randomized, single-arm study to assess the safety and efficacy of the CEM-Cage used with the CEM-Plate in patients who are appropriate candidates for a 2-level anterior cervical discectomy and fusion (ACDF). Fifty patients will be enrolled in the study and, after undergoing a 2-level ACDF, will be evaluated at 4 weeks, 3 months, 6 months, 12 months, 18 months, and 24 months.

The study consists of a screening period, surgical procedure, and 6 post-operative visits. At each indicated visit, quality of life scales and adverse events will be collected. In addition, at 4 weeks post-operatively, patients will undergo static lateral cervical plain x rays to assess implant positioning and integrity. At 3 months, 6 months, 12 months, 18 months, and 24 months, patients will undergo flexion/extension and neutral lateral plain radiographs to assess overall success and fusion.

The study has co-primary endpoints for efficacy (fusion) and overall success where overall success is defined as fusion, device implanted as intended, no serious adverse events related to the surgical procedure, no device-related serious adverse events, no subsequent surgical interventions at the index levels, and absence of clinically significant device malfunctions. Fusion data will be compared to benchmark data (Davis et al, 2013, control arm of the 2-level Mobi-C IDE study).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 22-79 years.
2. Documented diagnosis of cervical spine radiculopathy or myelopathy.
3. Symptomatic cervical degenerative disc disease at 2 contiguous levels between C2 through T1.
4. Baseline NDI score ≥30 and/or baseline mJOA score ≤16.
5. Pathology at the level to be treated correlating to the primary symptoms confirmed by imaging (computed tomography (CT), CT myelography, magnetic resonance imaging (MRI), or plain radiography).
6. Unresponsive to non-operative, conservative treatment for at least 6 weeks from symptom onset or presence of progressive cervical myelopathy or signs of nerve root/spinal cord compression despite continued non-operative treatment.
7. Ability to speak, read, and understand the IRB approved Informed Consent document.
8. Willingness to give informed consent for participation in the study.

Exclusion Criteria:

1. Any prior cervical surgeries at the symptomatic levels; prior surgery or cervical fusion procedure at any level.
2. Fewer than 2 or more than 2 vertebral levels requiring treatment.
3. Anatomy that is non-conducive to receiving investigational device.
4. More than one immobile vertebral level between C-1 to C-7 from any cause, including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions.
5. Known diagnosis of osteoporosis, current pharmacological treatment for osteoporosis or bone density which in the medical opinion of the surgeon precludes operation or contraindicates instrumentation.
6. Paget disease, osteomalacia, or any other metabolic bone disease other than osteoporosis.
7. Active malignancy that includes a history of any invasive malignancy (except nonmelanoma skin cancer), unless previously treated with curative intent and with no clinical signs or symptoms of the malignancy for > 5 years.
8. Severe cervical instability based on radiographic exam (whereby an anterior and posterior reconstructive procedure is indicated).
9. Decompression requiring corpectomy at one or more levels.
10. Active systemic infection or an infection localized to the site of the proposed implantation.
11. Open wounds.
12. Signs of local inflammation.
13. Fever.
14. Any diseases or conditions that would preclude accurate clinical evaluation.
15. Daily, high-dose oral and/or inhaled steroids or a history of chronic use of high-dose steroids.
16. BMI > 40.
17. Use of any other investigational drug or medical device within 30 days prior to surgery.
18. Smoking more than 1 pack of cigarettes/day.
19. Mental illness that, in the opinion of the investigator, would preclude patient's ability to participate in the study.
20. Current or recent history of substance abuse (alcoholism and/or narcotic addiction) requiring intervention.
21. Litigation relating to spinal injury/worker's compensation.
22. Reported to have a history of or anticipated treatment for active systemic infection, including human immunodeficiency virus (HIV) or Hepatitis C.
23. Previous trauma to the C2 to T1 levels resulting in significant bony or disco-ligamentous cervical spine injury.
24. Axial neck pain in the absence of other symptoms of radiculopathy or myeloradiculopathy or myelopathy justifying the need for surgical intervention.
25. Pregnancy.
26. Any medical or surgical condition which would preclude the potential benefit of spinal implant surgery, such as the elevation of sedimentation rate unexplained by other diseases, elevation of white blood count (WBC), or a marked left shift in the WBC differential count.
27. Suspected or documented metal allergy or intolerance.
28. Inadequate tissue coverage over the operative site or where there is inadequate bone stock, bone quality, or anatomical definition.
29. Any patient unwilling to cooperate with the post-operative instructions.
30. Any time implant utilization would interfere with anatomical structures or expected physiological performance.

Ages: 22 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-03-07 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Fusion | 24 months.
  Flexion-extension plain radiographs and CT scans will be used to assess bony fusion at both surgical levels.

SECONDARY OUTCOMES:
Device-Related Adverse Events | 24 months.
  No serious adverse events related to the surgical procedure, no device-related serious adverse events, no subsequent surgical interventions at the index levels, and absence of clinically significant device malfunctions.

CONTACTS AND LOCATIONS:
Overall Officials: John German, MD, Principal Investigator — Albany Medical College
Locations (4):
- United States (4):
  - IGEA, Union, New Jersey
  - Albany Medical College, Albany, New York
  - University at Buffalo Neurosurgery, Williamsville, New York
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No